CLINICAL TRIAL: NCT02586974
Title: Effects of Warmed, Humidified CO2 Insufflation on Body Core Temperature and Cytokine Response: Head-to-head Randomized Comparison Versus Standard Insufflation During Robot Assisted Radical Prostatectomy
Brief Title: Effects of Warmed, Humidified CO2 Insufflation on Body Core Temperature and Cytokine Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: IRCAD - EITS (Unknown)
Responsible Party: Principal Investigator, Marco Oderda, PhD fellow, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0052588
Record Dates: First submitted 2015-05-26; First posted 2015-10-27 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Hypothermia
Keywords: CO2 insufflation; robot assisted radical prostatectomy; laparoscopy; hypothermia; cytokine response
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group H+WB (Experimental): 32 patients will receive warmed, humidified CO2 insufflation with the Humigard® device, along with the hot air warming blanket used as a routine in our institution (forced air warming blanket at 38°C : Bear Hugger®)
  Interventions: Device: Humigard
- Group WB (No Intervention): 32 patients will receive standard CO2 insufflation, along with the hot air warming blanket used as a routine in our institution (forced air warming blanket at 38°C : Bear Hugger® and a standard insufflation with non-humidified, non-heated CO2)

INTERVENTIONS:
Device: Humigard — warmed and humidified CO2 insufflation
  Arms: Group H+WB

SUMMARY:
The aim of this study is to assess if the conditioning of the insufflation carbon dioxide (CO2) allows for an additional benefit in terms of prevention of the heat loss, when compared with the usual prevention with a forced warm air blanket alone, in the setting of robot-assisted radical prostatectomy (RARP).

DETAILED DESCRIPTION:
Among the possible consequences of cool and dry gas insufflation during laparoscopic procedures are hypothermia and cytokine response, which might cause significant perioperative morbidity. More in detail, body core temperature decrease during laparoscopic surgery has been calculated in humans as 0.3 °C for every 50 L of cold and dry insufflation gas. The reported temperature drop is caused by redistribution of heat and heat loss, both non-specific (due to anaesthesia and environmental patient exposure) and specific (due to peritoneal dry and cool insufflations). The resulting hypothermia can be severe, particularly after prolonged surgery. As for cytokine response, an increase of several pro-inflammatory cytokines has been described following the irritating effect of peritoneal CO2 insufflation.

That said, various devices of conditioning of the insufflating gas have been investigated to reduce the specific heat losses resulting from peritoneal insufflations, as well as to evaluate the inflammatory response. Previous studies conducted on animal models and clinical settings have suggested that warmed and humidified insufflation allows for an improved maintenance of body core temperature, a reduction in the degree of inflammatory response and an improved quality of postoperative course, compared with standard insufflating gas. These findings, however, are still not conclusive as they have not been confirmed by adequate randomized, controlled trials. Furthermore, no device providing warming and humidification has demonstrated a conclusive advantage over standard cold dry gas in terms of prevention of hypothermia during laparoscopy in man.

On the basis of the current available studies favouring warmed and humidified insufflation, the investigators hypothesize that a new device providing warmed and humidified insufflation (Humigard® Fisher and Paykel Healthcare®) might achieve significant benefits over standard insufflation in terms of body core temperature maintenance. The investigators also expect to document a decrease of pro-inflammatory cytokines, as a response to a diminished peritoneal irritation.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing RARP, with or without pelvic lymph node dissection, with a CO2 insufflation scheduled to last more than 60 minutes

Exclusion Criteria:

* patients over 80 years old, patients American Society of Anesthesiologist (ASA) status 4 or higher, patients not willing to sign the informed consent, conversions to open surgery

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gontero, Prof, Principal Investigator — AOU Città della Salute e della Scienza
Locations (1):
- A.O.U. San Giovanni Battista Molinette, Torino, TO, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients undergoing RARP at Città della Salute e della Scienza Hospital between September 2015 and June 2016 were screened for inclusion.
Pre-assignment Details: Exclusion criteria were as follows: age >80 years, ASA status >3, allergic status needing corticosteroid premedication, refusal to sign the informed consent, cognitive disability, conversion to open surgery.
Period: Overall Study
Arm/Group | Group H+WB | Group WB
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group H+WB | Group WB | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (7.0) | 64.4 (9.0) | 65.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 32 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 32 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Change in Body Core Temperature
Description: body core temperature of patients undergoing robot-assisted radical prostatectomy (RARP), measured with a disposable esophageal probe
Time Frame: Intraoperative at hourly intervals
Measure: Mean (Standard Deviation); unit: degrees °C
Groups:
- Group Humigard+Warming Blanket (H+WB): 32 patients will receive warmed, humidified CO2 insufflation with the Humigard® device, along with the hot air warming blanket used as a routine in our institution (forced air warming blanket at 38°C : Bear Hugger®)
  Humigard: warmed and humidified CO2 insufflation
- Group Warming Blanket (WB): 32 patients will receive standard CO2 insufflation, along with the hot air warming blanket used as a routine in our institution (forced air warming blanket at 38°C : Bear Hugger® and a standard insufflation with non-humidified, non-heated CO2)
Arm/Group | Group Humigard+Warming Blanket (H+WB) | Group Warming Blanket (WB)
Number analyzed (Participants) | 32 | 32
degrees °C
  start of surgery | 35.73 (0.37) | 35.70 (0.34)
  after 1h | 35.78 (0.42) | 35.77 (0.37)
  after 2h | 35.96 (0.53) | 35.90 (0.41)
  after 3h | 36.11 (0.60) | 36.07 (0.52)
  after 4h | 36.34 (0.64) | 36.07 (0.55)
  end of surgery | 36.26 (0.69) | 36.06 (0.62)

2. Secondary Outcome: Cytokine Interleukin-6 (IL-6)
Description: mean levels of the pro-inflammatory cytokine interleukin-6 (IL-6) in patients undergoing robot-assisted radical prostatectomy (RARP), measured just before induction of anesthesia, after 2 h of pneumoperitoneum, 2 h from exsufflation, and 24 h after surgery
Time Frame: changes in cytokine levels measured just before induction of anesthesia, after 2 h of pneumoperitoneum, 2 h from exsufflation, and 24 h after surgery
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Group H+WB | Group WB
Number analyzed (Participants) | 32 | 32
IU
  start of surgery | 2.13 (2.07) | 2.20 (2.2)
  after 2h | 4.61 (5.04) | 4.16 (3.5)
  2h from exsufflation | 29.13 (24.18) | 25.91 (22.9)
  24h after surgery | 27.01 (25.12) | 23.67 (25.8)

3. Secondary Outcome: Cytokine Tumor Necrosis Factor (TNF)-Beta
Description: mean levels of the pro-inflammatory cytokine tumor necrosis factor (TNF)-beta in patients undergoing robot-assisted radical prostatectomy (RARP), measured just before induction of anesthesia, after 2 h of pneumoperitoneum, 2 h from exsufflation, and 24 h after surgery
Time Frame: changes in cytokine levels just before induction of anesthesia, after 2 h of pneumoperitoneum, 2 h from exsufflation, and 24 h after surgery
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Group H+WB | Group WB
Number analyzed (Participants) | 32 | 32
IU
  start of surgery | 5.74 (4.8) | 6.29 (6.6)
  after 2h | 5.69 (5.8) | 5.20 (4.2)
  2h from exsufflation | 5.44 (5.3) | 4.90 (4.5)
  24h after surgery | 6.11 (5.7) | 7.24 (6.0)

4. Secondary Outcome: Postoperative Pain
Description: postoperative pain in patients undergoing robot-assisted radical prostatectomy (RARP) as measured by the Numeric Pain Rating Score (NRS), measured at patient awakening and after 12, 24, and 48 h from surgery. NRS goes from 0 to 10, where 0 means no pain and 10 the maximum pain possible.
Time Frame: changes in postoperative pain measured at patient awakening and then every 30 min in the recovery room, until discharge to the ward. Successively, it was measured at 12, 24, and 48 h
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group H+WB | Group WB
Number analyzed (Participants) | 32 | 32
Units on a scale
  Patient awakening | 2.5 (2.6) | 2.3 (2.8)
  At 12 hours | 1.6 (1.8) | 1.9 (2.2)
  At 24 hours | 1.3 (1.5) | 1.8 (2.1)
  At 48 hours | 0.6 (1.1) | 1.1 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse event data during hospital stay, an average of 4 days
Description: Adverse events (as per Clavien-Dindo classification) directly linked to the CO2 insufflation during the robot-assisted laparoscopic procedure (standard vs Humigard)
Arm/Group | Group H+WB | Group WB
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes